CLINICAL TRIAL: NCT02958683
Title: An Observational Study of Chest Wall Motion Analysis in Disease
Brief Title: Chest Wall Motion Analysis in Disease
Acronym: CWM
Status: Completed | Type: Observational
Sponsor: Heart of England NHS Trust (Other)
Collaborators: University of Birmingham (Other); University of Warwick (Other)
Responsible Party: Sponsor
Other Study IDs: 2010109TS
Record Dates: First submitted 2016-08-05; First posted 2016-11-08 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Mesothelioma; Lung Neoplasms; Surgery; Cystic Fibrosis; Pectus Carinatum; Pectus Excavatum; Empyema, Pleural; Pulmonary Disease, Chronic Obstructive
Keywords: Optoelectronic plethysmography; Structure light plethysmography; Respiratory Function Tests
MeSH Terms: conditions — Mesothelioma; Lung Neoplasms; Cystic Fibrosis; Pectus Carinatum; Funnel Chest; Empyema, Pleural; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (10):
- Pectus excavatum: Patients with pectus excavatum (funnel chest) condition undergo chest wall motion analysis
  Interventions: Other: Chest wall motion analysis
- Pectus carinatum: Patients with pectus carinatum (pigeon chest) condition undergo chest wall motion analysis
  Interventions: Other: Chest wall motion analysis
- Chronic obstructive pulmonary disease: Patients affected by COPD undergo chest wall motion analysis
  Interventions: Other: Chest wall motion analysis
- Diaphragm abnormality: Patients with abnormal function or structure of the diaphragm. Including diaphragmatic hernia/rupture and diaphragmatic paralysis undergo chest wall motion analysis
  Interventions: Other: Chest wall motion analysis
- Healthy control: People who do not have any diagnosed thoracic condition and who do not have symptoms/signs suggestive of undiagnosed thoracic disease undergo chest wall motion analysis
  Interventions: Other: Chest wall motion analysis
- Lung cancer: Patients with suspected or confirmed lung malignancy of all histological subtypes undergo chest wall motion analysis
  Interventions: Other: Chest wall motion analysis
- Pleural disease: Patients with pleural thickening and/or pleural effusion, pneumothorax, empyema undergo chest wall motion analysis
  Interventions: Other: Chest wall motion analysis
- Asthma: Patients diagnosed with asthma clinically or upon spirometry undergo chest wall motion analysis
  Interventions: Other: Chest wall motion analysis
- Cystic fibrosis: Patients diagnosed with cystic fibrosis clinically or biochemically undergo chest wall motion analysis
  Interventions: Other: Chest wall motion analysis
- Rib or sternal disease: Patients with an abnormality in the chest wall including fractures, osteomyelitis, malignancy of all histological subtypes, chest wall resection/reconstruction undergo chest wall motion analysis
  Interventions: Other: Chest wall motion analysis

INTERVENTIONS:
Other: Chest wall motion analysis — Assessment of chest wall motion using novel technologies including: optoelectronic plethysmography (OEP), structured light plethysmography (SLP), Microsoft Kinnect

SUMMARY:
Breathing movements, called chest wall motion, are very complex. The investigators are studying how movement of the abdomen, ribs and diaphragm contribute to breathing and how this differs with different diseases in the chest. Breathing movements may help with diagnosis, assessment of severity or assessing the impact of treatments for chest conditions. The investigators are following people who have a chest disease, measuring their chest wall motion and comparing it to their diagnosis and and how their treatment works.

Chest wall motion can be measured in different ways at rest and whilst exercising. Small stickers on the chest can be used to reflect infra red light or visible squares of light can be shone onto the chest without using stickers.

DETAILED DESCRIPTION:
Optoelectronic plethysmography (OEP) is based on the analysis during breathing of the trajectories of a series of markers positioned on the thoracic-abdominal surface of the patient. The positions in space of these markers are recorded and processed with mathematical models and algorithms by a computing unit that can accurately measure not only volume variations of the whole thoracic-abdominal wall, but also the variations of the various compartments. This detects, for example, asymmetries in the action of respiratory muscles. The system can accurately measure current volume, vital capacity, respiratory frequency, duration of the phases of inspiration and exhalation, the average inspiration and exhalation flux and the volume variations at the end of exhalation.

Structured Light Plethysmography (SLP) also assesses regional chest wall excursion but does not require markers to be placed on the patient. The system uses visible light shone onto the chest wall in a checkerboard pattern and reflected back by the patient's skin or a tight T shirt.

Images from 4 Microsoft Kinnect Motion Cameras can be used to create a 3D representation of the patient's torso. This system has been shown to correlate well with chest wall measurements recorded by OEP.

These systems are innovative examination instruments, non-invasive, accurate, easy to use and unlike traditional plethysmographic technologies, are not affected by humidity and temperature variations and can easily be used to perform measurements for extended periods of time. They accurately measure the dynamics of the volume variations that occur during breathing in the various sections of the thoracic-abdominal walls (upper, lower and abdominal thoracic area). This data, which is otherwise undetectable, is a useful contribution to the evaluation of patients. We will apply chest wall motion analysis to understanding the physiology of thoracic disease processes as well as assessing potential diagnostic and prognostic (response to treatment) markers that could be used in future clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16 or over
* Have thoracic disease or healthy control

Exclusion Criteria:

* Unable to provide valid informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients or their healthy acquaintances attending Heart of England NHS Foundation trust for care under the thoracic surgery department or respiratory department.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2011-07 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2015-07-31 (Actual)

PRIMARY OUTCOMES:
Change in volume of each thoracoabdominal compartment during breathing | Baseline, follow up after normal clinical care up to 3 times (inpatient after surgery, 4-6 weeks, 3-12 months)
  Measured in litres

SECONDARY OUTCOMES:
Synchrony of chest wall movement | Baseline, follow up after normal clinical care up to 3 times (inpatient after surgery, 4-6 weeks, 3-12 months)
  Measured in degrees

CONTACTS AND LOCATIONS:
Overall Officials: Babu Naidu, MBBS, Principal Investigator — Heart of England NHS Foundation Trust
Locations (1):
- Heart of England NHS Foundation Trust, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aliverti A, Pedotti A. Opto-electronic plethysmography. Monaldi Arch Chest Dis. 2003 Jan-Mar;59(1):12-6. PMID 14533277
- [Derived] Oswald N, Jalal Z, Kadiri S, Naidu B. Changes in chest wall motion with removal of Nuss bar in repaired pectus excavatum - a cohort study. J Cardiothorac Surg. 2019 Jan 8;14(1):4. doi: 10.1186/s13019-018-0827-1. PMID 30621729